CLINICAL TRIAL: NCT00247572
Title: A Double-Blind Placebo- and Active-Controlled, Single-Dose Crossover PD and PK Study to Evaluate the Safety, Tolerability and Abuse Liability of IV Administered NRP104 25 mg and 50 mg in Adult Volunteers With Histories of Stimulant Abuse
Brief Title: Safety, Tolerability and Abuse Liability Study of Intravenous NRP104 in Adults With Stimulant Abuse Histories
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New River Pharmaceuticals (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NRP104.A02; WIRB(R) Protocol #20051316
Record Dates: First submitted 2005-10-31; First posted 2005-11-02 (Estimated); Last update posted 2007-11-05 (Estimated); Status verified 2007-11

CONDITIONS: Attention Deficit Disorder With Hyperactivity; Amphetamine-Related Disorders; Substance-Related Disorders
Keywords: d-Amphetamine; Attention Deficit Hyperactivity Disorder; Attention Deficit Disorders with Hyperactivity; Attention Deficit Hyperactivity Disorders; Amphetamine Abuse; Amphetamine Dependence; Amphetamine Addiction; Amphetamine Users; Drug Abuse; Drug Addiction; Drug Dependence; Drug Habituation; Drug Use Disorders; Substance Abuse; Substance Dependence; Substance Use Disorders; Drug Usage; Substance Addiction; Drug Abuse, Intravenous; Intravenous Drug Abuse
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Amphetamine-Related Disorders; Substance-Related Disorders; Substance Abuse, Intravenous | interventions — Lisdexamfetamine Dimesylate

INTERVENTIONS:
Drug: NRP104

SUMMARY:
This research is being done to evaluate if NRP 104 is a safe drug. The other purpose is to learn if NRP104, when injected into a vein, produces a high and any other effects like amphetamine and other stimulant drugs that are abused. This information will give some indication if NRP104 can be abused. Healthy people, between the ages of 18 and 55 with histories of substance abuse that include stimulant drugs, may join. Amphetamines are drugs that are used most often to treat attention deficit hyperactivity disorder (ADHD) in children, to treat narcolepsy (excessive sleepiness) and for weight loss.

DETAILED DESCRIPTION:
There is a need for a non-scheduled stimulant medication that can provide symptom control for children with ADHD as the conventional stimulant products do.

Currently, the top line amphetamine product Adderall XR (R) for the treatment of children with ADHD involves a once-a-day morning dosing of up to 30 mg per day per Adderall XR (R) Package Insert. New River Pharmaceuticals has developed three NRP104 dose strengths of 30 mg, 50 mg, and 70 mg to provide amphetamine base equivalent to Adderall XR (R) 10 mg, 20 mg, and 30 mg, respectively. Adderall XR (R) and other amphetamine and methylphenidate containing preparations are liable to intravenous abuse.

As part of the development of NRP104 for treatment of children with ADHD, it is important to evaluate the abuse potential of NRP104 given intravenously in comparison to immediate release d-amphetamine. This study will conduct relevant information to address appropriately the objectives of determining abuse potential of intravenously administered NRP104.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject is 18 to 55 years of age, inclusive.
* Except for women who are post menopausal or surgically sterile, all female subjects must have a negative urine pregnancy test at screening and at admission to the research unit. They must abstain from sexual activity, or use acceptable contraceptives throughout the study, and for 30 days after the last dose of study drug. Acceptable contraceptives include double barrier method (such as condom with spermicidal gel or diaphragm with spermicidal gel), IUDs and hormonal contraceptives which must be pharmacologically effective prior to study drug exposure.
* Meet DSM-IV criteria for the diagnosis of substance abuse.
* Have a history of IV drug use.
* Subject must be in good health and have venous access sufficient for (1) IV drug administration and (2) blood collection, as determined by medical history, physical exam, and clinical labs.
* Agree to be admitted to the inpatient research unit for a minimum of 8 days, and be able to complete all protocol-specified assessments.
* Able to understand that they can withdraw from the study at any time.
* Minimum reading level of Grade Six as determined by the REALM test, at the investigator's discretion.
* Subject must voluntarily consent to participate in this study.

Exclusion Criteria:

* History of clinically significant gastrointestinal, renal, hepatic, endocrine, oncologic, hematologic, neurologic, psychologic, immunologic or pulmonary disorders; or cardiovascular disease, tuberculosis, epilepsy, diabetes, psychosis, glaucoma, or any condition which in the opinion of the Investigator would jeopardize the safety of the subject or impact study results or prevent the subject from completing the study.
* Presence or history of any medically diagnosed, clinically significant Axis I psychiatric disorders other than substance abuse (including bipolar disorder, any psychotic disorder, and Tourette's disorder or family history of Tourette's).
* Serious suicidal risk determined by the investigator.
* Presence of a severe learning difficulty or mental retardation, or any condition that would interfere with participation or completion of the study.
* History of allergic or adverse response or hypersensitivity to d-amphetamine or NRP104.
* Participation in a previous clinical trial within 30 days prior to study initiation.
* Blood loss, donation of one pint or more, or plasma donation within 60 days prior to study initiation.
* Clinically significant abnormalities at screening or admission on results of ECG or lab tests, including lab deviations requiring acute medical intervention or further medical attention.
* Treated with a monoamine oxidase inhibitor, currently or within 13 days of initiation of the study medication.
* Require any of the following medications: clonidine or other alpha-2 adrenergic receptor agonists, tricyclic antidepressants, selective serotonin reuptake inhibitors (SSRIs) theophylline, coumarin anticoagulants, or anticonvulsants; or have taken an SSRI in the 35 days before initiation of the study medication.
* Currently physically dependent on benzodiazepines as determined by clinical evaluation and/or urine drug screen at screening.
* Currently physically dependent on opiates as determined by naloxone challenge.
* Currently physically dependent on alcohol as determined by clinical evaluation or has a positive Breathalyzer test at screening or admission and confirmed by a second reading.
* Preexisting severe gastrointestinal narrowing.
* Use of any prescription medications (except birth control methods) within 14 days of admission, or will require any prescription medications, or any over-the-counter (OTC) medications (other than acetaminophen), or herbal supplements or vitamins during the study.
* Positive urine pregnancy test at screening or admission.
* Female subject is pregnant or lactating.
* Another member of the subject's household currently participating in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2005-09; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic (PD) Parameters:
The following parameters will be measured at fixed time intervals post drug and used to compare the
effects of various doses of NRP104 with placebo and d-amphetamine sulfate for pharmacodynamic
equivalence:
(1) Maximum liking scale scores for euphoria measured by DRQS and DRQO
(2) Maximum disliking scale scores for dysphoria measured by DRQS and DRQO
(3) Maximum scores on the MBG, BG and Amphetamine scales of the ARCI
(4) Maximum supine systolic and diastolic blood pressure changes from baseline
(5) Maximum orthostatic pulse increases from baseline
(6) Spontaneous reports of discomforting subjective effects
(7) Adverse events, laboratory tests, physical examination, vital signs and ECG will be collected to
assess the safety and tolerability of NRP104.
Pharmacokinetic (PK) Parameters
The following parameters will be calculated using non-compartmental analysis for d-amphetamine and
intact
NRP104: AUC0-24, Cmax , Tmax.
• AUC0-24: Area under the drug concentration-time curve from time zero to 24 hours post dose.
• Cmax: Maximum observed drug concentration from zero hour to 24 hours post dose.
• Tmax: Time at which Cmax occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Jasinski, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Clinical Studies Program, Baltimore, Maryland, United States